CLINICAL TRIAL: NCT02496598
Title: In Vitro Activation of Primordial Follicles as a Method to Treat Infertility Caused by Primary Ovarian Insufficiency
Brief Title: In Vitro Follicle Activation
Acronym: IVA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results were not promising
Sponsor: National Foundation for Fertility Research (Other)
Collaborators: Fertility Laboratories Of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFFR-IVA-2015
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Primary Ovarian Insufficiency; Infertility
Keywords: Reproductive Techniques, Assisted; Ovarian Follicle
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility; Helping Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- In Vitro Follicle Activation (IVA) (Experimental): Ovarian tissue will be removed and cultured in vitro with compounds to activate dormant follicles. Following activation, ovarian tissue will be auto-grafted and the patient monitored for follicular growth.
  Interventions: Procedure: In Vitro Follicle Activation (IVA); Drug: Follicle Activation

INTERVENTIONS:
Procedure: In Vitro Follicle Activation (IVA) — Laparoscopic removal of ovarian tissue, followed by in vitro activation of dormant ovarian follicles and autografting back to the patient for follicle growth and egg retrieval.
Drug: Follicle Activation — Ovarian cortical pieces will be treated in vitro with a PTEN activator (bpV(hopic)) and a PI3K inhibitor (740YP) in vitro to activate primordial ovarian follicles, prior to autografting.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an experimental treatment, known as in vitro activation (IVA) of dormant ovarian follicles, for infertility in women diagnosed with primary ovarian insufficiency (POI).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of an experimental treatment, known as in vitro activation (IVA) of dormant ovarian follicles, for infertility in women diagnosed with primary ovarian insufficiency (POI; also known as premature ovarian failure). Patients diagnosed with POI are infertile due to a lack of follicle growth and ovulation; oocyte donation is the only treatment option currently available to enable these women to have a child. IVA treatment may result in the rescue of the remaining primordial follicles within the ovary, thus making oocytes available for IVF, embryo production, transfer and pregnancy. In this experimental treatment, ovarian tissue is removed from the patient and cultured in vitro for 48 hours with specific compounds to activate dormant primordial follicles. Following activation ovarian tissue is auto-grafted to the serosa of the fallopian tube, and the patient is monitored for signs of follicle growth. Growing follicles are stimulated with exogenous hormones, followed by oocyte retrieval and IVF.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with primary ovarian insufficiency (POI), seeking pregnancy and eligible for IVF at Colorado Center for Reproductive Medicine (Lone Tree, CO).
* Patients can be of any race, culture, sexual orientation or ethnicity.

Exclusion Criteria:

* Minors are excluded from participation in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Antral follicle development measured by ultrasound examination | 1 year after auto-grafting
  Ultrasound analysis of the number of follicles developing in the grafted ovarian tissue following activation in vitro
Recovery of oocytes by trans-vaginal ultrasound guided oocyte aspiration | 1 year after auto-grafting
  The number of oocytes recovered from follicles developing in the grafted ovarian tissue following in vitro activation
Pregnancy | 1.5 years after auto-grafting
  The incidence of implantation and pregnancy following transfer of embryos produced from oocytes recovered from follicles developing in the activated ovarian tissue.

SECONDARY OUTCOMES:
Offspring weight | 1 year after egg retrieval
  The birth weight of children born
Offspring gender | 1 year after egg retrieval
  The gender of children born
Development of good quality blastocysts using the Gardner morphological blastocyst grading system | 1 week after egg retrieval
  The proportion of good quality blastocyst stage embryos developed during in vitro fertilization (IVF) cycle(s), of the total number of fertilized eggs

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Krisher, Ph.D., Principal Investigator — NFFR; William B Schoolcraft, M.D., Principal Investigator — Fertility Laboratories Of Colorado
Locations (2):
- United States (2):
  - Fertility Laboratories of Colorado, Lone Tree, Colorado
  - National Foundation for Fertility Research, Lone Tree, Colorado

REFERENCES:
- [Background] Kawamura K, Cheng Y, Suzuki N, Deguchi M, Sato Y, Takae S, Ho CH, Kawamura N, Tamura M, Hashimoto S, Sugishita Y, Morimoto Y, Hosoi Y, Yoshioka N, Ishizuka B, Hsueh AJ. Hippo signaling disruption and Akt stimulation of ovarian follicles for infertility treatment. Proc Natl Acad Sci U S A. 2013 Oct 22;110(43):17474-9. doi: 10.1073/pnas.1312830110. Epub 2013 Sep 30. PMID 24082083
- [Background] Suzuki N, Yoshioka N, Takae S, Sugishita Y, Tamura M, Hashimoto S, Morimoto Y, Kawamura K. Successful fertility preservation following ovarian tissue vitrification in patients with primary ovarian insufficiency. Hum Reprod. 2015 Mar;30(3):608-15. doi: 10.1093/humrep/deu353. Epub 2015 Jan 6. PMID 25567618